CLINICAL TRIAL: NCT02839135
Title: A Randomized, Single-center, Crossover, Comparative Bioavailability and Adhesion Performance Study, Comparing Single Administrations of a New Scopolamine Transdermal Delivery System Formulation to the Currently Established Reference Transdermal Delivery System in Healthy Adult Participants.
Brief Title: A Comparative Bioavailability and Adhesion Performance Study, Comparing a New Scopolamine Transdermal Delivery System Formulation to the Currently Established Reference Transdermal Delivery System in Healthy Adult Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 205035
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Reformulated scopolamine patch (Experimental): Participants will receive reformulated scopolamine Transdermal Delivery System (TDS) patch 1.5 mg (+/- 0.3 mg) /system of 2.5 cm2 surface area with delivery of approximately 1.0 mg over 72 hours.
  Interventions: Drug: Reformulated scopolamine patch
- Marketed scopolamine patch (Active Comparator): Participants will receive currently marketed scopolamine TDS patch 1.5 mg (+/- 0.3 mg) /system of 2.5 cm2 surface area, with delivery of approximately 1.0 mg over 72 hours.
  Interventions: Drug: Marketed scopolamine patch

INTERVENTIONS:
Drug: Reformulated scopolamine patch — Reformulated scopolamine patch of 1.5 mg (+/- 0.3 mg) /system of 2.5 cm2 surface area with deliver approximately 1.0 mg over 72 hours
  Arms: Reformulated scopolamine patch
Drug: Marketed scopolamine patch — Marketed scopolamine patch of 1.5 mg (+/- 0.3 mg) /system of 2.5 cm2 surface area with delivery of approximately 1.0 mg over 72 hours.
  Arms: Marketed scopolamine patch

SUMMARY:
In this comparative bioavailability and in vivo skin adhesion study, the impact of minor changes in qualitative composition of polyiso-Butylenes (PIB) from a different supplier and change of the manufacturing line of the micro porous membrane will be tested.

DETAILED DESCRIPTION:
This study is a randomized, single-center, cross-over, comparative bioavailability and adhesion study, comparing single administrations of a new scopolamine transdermal delivery system formulation to the current established reference transdermal delivery system in healthy adult participants. The study will consist of an ambulant screening day within 21 days prior to the first investigational medicinal product (IMP) administration at study Day 1 and two treatment periods. Each treatment period will consist of 4.5 days (108 hours) of in-house confinement.

ELIGIBILITY:
Inclusion Criteria:

* Participants must understand and provide written informed consent before any assessment is performed, understand the study procedures, and be willing and able to complete the required assessments.
* Male or female participants of any ethnic origin, and aged from 18 to 55 years (inclusive).
* Body mass index between 18 and 30 kg/m2.
* Normal vital signs as follows: Oral body temperature between 35.0 and 37.5 ºC (95 and 99.5 °F) inclusive; Supine systolic blood pressure between 90 and 140 mmHg inclusive; Supine diastolic blood pressure between 55 and 90 mmHg inclusive;Pulse rate between 50 and 100 beats per minute (bpm) inclusive.
* In general good physical health including the presence of healthy and non irritated skin at test site behind the participant's ears, as judged by the investigator and determined by medical/surgical history, physical examination, electrocardiogram (ECG) (12-lead), and clinical laboratory (clinical chemistry, hematology and urinalysis).
* Ability to communicate and comply with all study requirements.
* Willingness and ability to complete the study.

Exclusion Criteria:

* Presence of tattoo, hair (including shaved hair) or scarring on the test site behind the participant's left or right ear.
* Surgical procedures or use of topical pharmacologic treatments directly over the test site(s) within 90 days before enrollment.
* Use of other belladonna alkaloids, antihistamines, tricyclic antidepressants (such as amitriptyline and imipramine), amantadine, quinidine within 2 weeks prior to the first scheduled study drug administration.
* Participation in a previous clinical study with another investigational product within the last 90 days or use of other investigational drugs within 90 days or 10 half-lives before enrollment, whichever is longer.
* History of or known hypersensitivity or photosensitivity to any of the study drugs, excipients or to drugs of similar chemical classes.
* Diagnosis of angle-closure (narrow angle) glaucoma.
* History or current evidence of pyloric obstruction, intestinal obstructions or urinary bladder neck obstruction (e.g. due to benign prostate hyperplasia) and History of seizures or psychosis.
* Diagnosis of long QT syndrome or QTc > 450 millisecond (msec) for males and > 470 msec for females at screening.
* History of malignancy or neoplastic disease of any organ system (except for localized basal cell skin carcinoma), treated or untreated, within the past 5 years prior to screening, regardless of whether there is evidence of local recurrence or metastases.
* Pregnant, nursing (lactating) women.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant unless they are: women whose career, lifestyle or sexual orientation precludes intercourse with a male partner, at the judgment of the investigator; women who have been surgically sterilized or whose partners have been sterilized by vasectomy or other means; using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices (IUDs). Double barrier and periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) are not acceptable means of contraception; A woman who is postmenopausal must have a negative urine pregnancy test at screening but will not need to comply with an acceptable method of contraception. Women are considered post-menopausal and not of child bearing potential if they had 12 months of natural (sp ntaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with known or reported serum FSH levels > 40 mIU/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks before. In the case of oophorectomy alone, women are considered post-menopausal only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance.
* History of hypertension, cardiovascular disease, stroke or Transient Ischemic Attack (TIA).
* History of orthostatic hypotension, fainting or blackouts.
* Clinically relevant chronic or acute infectious illnesses or febrile infections within two weeks prior to start of the study.
* History within the last five years or current evidence of pulmonary, gastrointestinal, hematological, endocrinological, metabolic, autoimmune, neurological, psychiatric or other diseases at screening unless deemed medically insignificant or clinically insignificant as assessed by the Investigator.
* Clinically significant laboratory findings at screening such as anemia (hemoglobin <11.5 g/dL for women and <13.5 g/dL for men), serum potassium <3.5 mmol/L or >5.0 mmol/L, or serum sodium <132 mmol/L or >150 mmol/L.
* Use of any medication within 2 weeks before first scheduled study drug administration or within less than 10 times the elimination half-life of the respective drug (whichever is longer), or is anticipated to require any concomitant medication during that period or at any time throughout the study.
* Any history of asthma, urticaria, or other significant allergic diathesis. Participants with uncomplicated seasonal allergic rhinitis can be accepted if expected allergy season is clearly outside enrolment/ treatment period.
* Participant has a history of illicit drug abuse or investigator has evidence of current drug abuse with drug classes that include but are not limited to barbiturates, tricyclic antidepressants, amphetamines, benzodiazepines, cocaine, opiates, cannabis or any other illicit drugs (verified by urine drug screen or other reliable evidence).
* Smokers or evidence for current alcohol abuse or reports a regular average alcohol consumption exceeding 18 g (women) or 35 g (men) of pure alcohol per day, i.e. 1 drink/day for women or or 35 g (men) of pure alcohol per day, i.e. 1 drink/day for women or 2 drinks/day for men (1 drink = 5 oz of wine or 12 oz of beer or 1.5 oz of hard liquor) within 6 months of screening.
* Positive results in any of the virology tests for Human Immunodeficiency Virus Antibodies (HIV-Ab), Antibodies Hepatitis C Virus (HCV-Ab), Surface antigen of Hepatitis B (HBsAg) and HBc-Ab (Immunoglobulin G [IgG] +Immunoglobulin M [IgM]).
* Performance of unaccustomed strenuous physical exercise (body building, high performance sports) from 2 weeks prior to start of the study and throughout the entire study.
* Allergy to skin disinfecting agents, tape, or latex rubber.
* Any condition not identified in the protocol that in the opinion of the Investigator would confound the evaluation and interpretation of the study data or may put the participant at risk.
* Previously enrolled in the current study.
* "Vulnerable" individual.
* Participation in a clinical trial with at least 470mL blood drawn, or blood donation within 12 weeks prior to the start of the study.
* Not willing to fully comply with the following lifestyle restrictions throughout the study.
* Participation in a clinical trial with at least 470mL blood drawn, or blood donation within 12 weeks prior to the start of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-10 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | upto 96 hours
  The maximum observed post-dose concentration.
Area under the curve from time zero extrapolated to infinity [AUC(0-inf)] | upto 96 hours
  The area under the plasma concentration versus time curve will be calculated from time 0 to infinity.
Area under the curve from time zero to last sampling time [AUC(0-t)] | upto 96 hours
  The area under the plasma concentration versus time curve will be calculated from time 0 to the last measurable sampling time point, t.
Time to reach maximum plasma concentration (Tmax) | upto 96 hours
  The time of the maximum observed post-dose concentration.
Termination rate constant (Lambda_z) | upto 96 hours
  The terminal elimination rate constant.
Percentage area under the curve by extrapolation (%AUCex) | upto 96 hours
  Percentage of AUC0-inf obtained by extrapolation.
Elimination half life (t1/2) | upto 96 hours
  The elimination half-life.
Patch adherence assessment | upto Day 4
  Patch adherence evaluation will be performed.

SECONDARY OUTCOMES:
Skin Irritation | After 0.5 hour, 24 hours
  Skin irritation will be assessed at 0.5 hour and 24 hours after patch removal in each study period.
Safety Assessment | upto Day 16
  Safety assessments will consist of evaluation of skin for irritation, monitoring and recording of all adverse events including serious adverse events, physical examination, vital signs (including blood pressure, pulse rate and body temperature), laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mont Royal, QC, Quebec, Canada

REFERENCES:
- See also: Results for Study 205035 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/205035?search=study&study_ids=205035#rs